CLINICAL TRIAL: NCT00097643
Title: Problem Solving/Physical Interventions and Aging
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Linda Teri, PhD, Northwest Research Group on Aging, University of Washington School of Nursing
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: AG0009; 5R01AG014777-05 (NIH)
Record Dates: First submitted 2004-11-24; First posted 2004-11-25 (Estimated); Last update posted 2008-08-13 (Estimated); Status verified 2008-08

CONDITIONS: Aging
Keywords: exercise; health promotion; independent living; affective aspects
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Health Promotion

INTERVENTIONS:
Behavioral: exercise
Behavioral: health promotion

SUMMARY:
The purpose of this study is to examine the relative and combined efficacy of a physical activity and health promotion program to help sedentary adults over age 70 maintain an independent life style.

DETAILED DESCRIPTION:
The study recruited 273 participants from a community-based HMO for whom computerized health service utilization and cost data were already available, as well as cognitive, functional, and health status measures. The participants were randomly placed into one of four treatment groups: exercise, health promotion, combination exercise and health promotion, and routine medical care. Assessments for physical performance, emotional well-being, and physical and emotional health status were conducted at screening, baseline, after 3 months (post-treatment), and at 6, 12, and 18-month follow-up by interviewers blind to treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

* age 70 or older
* live independently
* less than 150 minutes regular exercise per week
* able to walk across a room without a person assisting
* English speaking
* planning to stay in local area for at least 6 months (duration of active study)

Exclusion Criteria:

* cancer
* heart attack
* stroke
* uncontrolled arrhythmia
* uncontrolled hypertension
* uncontrolled diabetes
* surgery during the past year
* ongoing mental health or psychiatric condition

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 273
Dates: Start 2000-09; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
physical health and function | screening, baseline, 3, 6, 12, and 18 months
affective status | screening, baseline, 3, 6, 12, and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Linda Teri, PhD, Principal Investigator — University of Washington School of Nursing, Northwest Research Group on Aging

REFERENCES:
- [Background] Seeman TE, Charpentier PA, Berkman LF, Tinetti ME, Guralnik JM, Albert M, Blazer D, Rowe JW. Predicting changes in physical performance in a high-functioning elderly cohort: MacArthur studies of successful aging. J Gerontol. 1994 May;49(3):M97-108. doi: 10.1093/geronj/49.3.m97. PMID 8169338
- [Background] Schulz R, Heckhausen J. A life span model of successful aging. Am Psychol. 1996 Jul;51(7):702-14. doi: 10.1037//0003-066x.51.7.702. PMID 8694390
- [Background] Strawbridge WJ, Cohen RD, Shema SJ, Kaplan GA. Successful aging: predictors and associated activities. Am J Epidemiol. 1996 Jul 15;144(2):135-41. doi: 10.1093/oxfordjournals.aje.a008900. PMID 8678044
- [Background] Stuck AE, Walthert JM, Nikolaus T, Bula CJ, Hohmann C, Beck JC. Risk factors for functional status decline in community-living elderly people: a systematic literature review. Soc Sci Med. 1999 Feb;48(4):445-69. doi: 10.1016/s0277-9536(98)00370-0. PMID 10075171
- [Background] King AC, Pruitt LA, Phillips W, Oka R, Rodenburg A, Haskell WL. Comparative effects of two physical activity programs on measured and perceived physical functioning and other health-related quality of life outcomes in older adults. J Gerontol A Biol Sci Med Sci. 2000 Feb;55(2):M74-83. doi: 10.1093/gerona/55.2.m74. PMID 10737689
- [Background] Nelson ME, Layne JE, Bernstein MJ, Nuernberger A, Castaneda C, Kaliton D, Hausdorff J, Judge JO, Buchner DM, Roubenoff R, Fiatarone Singh MA. The effects of multidimensional home-based exercise on functional performance in elderly people. J Gerontol A Biol Sci Med Sci. 2004 Feb;59(2):154-60. doi: 10.1093/gerona/59.2.m154. PMID 14999030
- [Background] Strawbridge WJ, Deleger S, Roberts RE, Kaplan GA. Physical activity reduces the risk of subsequent depression for older adults. Am J Epidemiol. 2002 Aug 15;156(4):328-34. doi: 10.1093/aje/kwf047. PMID 12181102